CLINICAL TRIAL: NCT01172743
Title: Collection of Blood for Gene Expression/Genomic Studies in Individuals With Diabetes (Qatar)
Status: Terminated | Type: Observational
Why Stopped: Lack of funding.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other); Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 0904010340; HMC Protocol # 9093/09 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes; Type-2; Adult Onset
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA will be extracted, and genome wide SNP analysis and promoter sequences for genes will be obtained. The goal is to find single nucleotide polymorphims (SNP), small changes in single genes that affect disease risk, to see if they correlate with diabetes. Serum will be stored for future studies, for a period of 6 years, to look at levels of proteins. Subjects who consent to participate in this study will have their serum stored for up to 6 years, inorder to be used for future studies on genomics.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes: Individuals with diabetes that fit eligibility criteria.
- Normal Control: Individuals without history of diabetes.

SUMMARY:
This protocol is designed to gather a small amount of blood for extraction of DNA for the study of the genetic basis of diabetes. The study population will include individuals with known diabetes, and controls without diabetes. Investigators aim to understand the genetics of diabetes, and will use the cells and serum from this blood to perform genotyping and gene expression studies of individuals with diabetes and relevant controls.

DETAILED DESCRIPTION:
This protocol is designed to collect a small amount of blood for extraction of DNA (genetic material) for the study of the genetic basis of diabetes. The study population will include individuals with known diabetes and controls without diabetes. Additionally, this protocol will recruit individuals from the following locations: the Qatar Diabetes Association, the governmental ministries of Qatar, and subjects who have participated in Dr. Bener's HMC protocol #231 entitled "A preliminary study of genetic pre-disposition to diabetic mellitus in the state of Qatar." Individuals with diabetes may also be recruited from the Hamad Hospital outpatient adult diabetes clinics (there are eight diabetes clinics each week) and/or from the population of subjects who previously participated in Dr. Mushlin's IRB approved protocol #0608008703 entitled "Comparing the Clinical Management and Genetic Markers of Diabetes in Qatar to International Standards" at Hamad Medical Corporation or IRB approved protocol #0602008388 entitled "The Impact of Cardiac and Genetic Risk Factors on Acute Myocardial Infarction and Cerebrovascular Stroke in Qatar: A Case-Control Study". In this protocol, researchers will survey medical records of patients with diabetes, in order to study the clinical characteristics of these individuals, and the researchers will collect blood to evaluate the genetic characteristics of individuals with diabetes. The researchers will also collect blood samples of individuals without diabetes to serve as control.

ELIGIBILITY:
Diabetes group

Inclusion criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Documented evidence of diabetes using at least one of the following: (1) blood tests consistent with Type-II diabetes; (2) oral glucose tolerance tests consistent with Type-II diabetes; (3) subject taking medication to treat Type-II diabetes.

Exclusion criteria:

* Individual refuses consent
* Pregnant females with gestational diabetes
* Type-I diabetes

Normal control group

Inclusion Criteria:

* Must provide informed consent
* Males or females ages 18 years and older
* Resolved gestational diabetes

Exclusion Criteria:

* Individual refuses consent.
* Individuals with history of diabetes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetes group will be taken from (1)individuals visiting the Medicine Department at the Hamad Medical Corporation(HMC), Qatar for standard clinical care, (2)outpatient adult individuals seen at the HMCdiabetes clinics, (3)individuals who have participated in the following IRB protocol #s:0608008703, #0602008388 and HMC protocol #231, (4)ndividuals who attend clinics at the Qatar Diabetes Association (QDA), and (5)Individuals who work at the governmental ministries of Qatar. Controls will be obtained from volunteers without a history of diabetes. Family members of patients may be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2009-06; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Study Director — Weill Cornell Medical College, NY and Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided